CLINICAL TRIAL: NCT06872749
Title: Effect on an Experimental Gel Containing Copaiba Oil-resin in the Control of Dentin Hypersensitivity: a Randomized Clinical Study
Brief Title: Effect of an Experimental Gel Containing Copaiba Oil-resin in the Control of Dentin Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Professor of the Graduate Program in Dentistry at the Federal University of Pará, Universidade Federal do Para
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6.787.218
Record Dates: First submitted 2025-01-16; First posted 2025-03-12 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-03

CONDITIONS: Pain; Dentin Sensitivity; Dentin Desensitizing Agents
MeSH Terms: conditions — Pain; Dentin Sensitivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo gel (Placebo Comparator): the group will receive the application of gel without active ingredient
  Interventions: Other: Placebo gel
- KF2 (Potassium nitrate gel) (Active Comparator): the group will receive the application of gel containing potassium nitrate
  Interventions: Other: KF2 (Potassium nitrate gel)
- Copaiba gel (Experimental): the group will receive the application of gel containing copaiba
  Interventions: Other: experimental Copaiba gel

INTERVENTIONS:
Other: Placebo gel — will receive the application of a placebo gel (without active ingredient), under the same conditions described for the experimental gel.
  Arms: Placebo gel
Other: KF2 (Potassium nitrate gel) — will receive application of potassium nitrate gel on hypersensitive dental surfaces, in an active way, for 10 minutes.
  Arms: KF2 (Potassium nitrate gel)
Other: experimental Copaiba gel — will receive the application of the experimental desensitizing gel on the vestibular surfaces of the hypersensitive teeth in an active manner, for 10 minutes.
  Arms: Copaiba gel

SUMMARY:
This randomized, single-blind, placebo-controlled clinical trial aims to clinically evaluate the effect of an experimental gel containing copaiba oleo-resin in the control of dentin hypersensitivity (DH) in non-carious cervical lesions (NCCL). Seventy-five hypersensitive teeth will be selected into three groups (N=25) and approved in three treatment sessions. The groups will be: GROUP P= water-soluble placebo gel without active ingredient; GROUP KF2: Potassium nitrate 5% + Sodium fluoride 2%; GROUP GC: Gel containing copaiba oleo-resin. A visual analogue scale (VAS) will be used to compare the DH after tactile stimulation with an exploratory probe and evaporative stimulation with air jets. The DH assessments will be performed at four times: baseline, after 1 week, 15 days and 30 days after the beginning of treatment.

DETAILED DESCRIPTION:
The sequence of application of the gels, whether active or placebo, will be as follows:

A professional prophylaxis will be performed using a rubber cup on the dental elements. The corresponding gel for each group will be applied with the aid of a micro-applicator and will remain undisturbed on the surface for 10 minutes. After the gel application time has elapsed, and while it is still on the teeth, the product will be rubbed with a micro-applicator using circular and intermittent movements. Subsequently, the gel will be removed with cotton and abundant water.

ELIGIBILITY:
Inclusion Criteria:

* hypersensitive areas on the vestibular surface of the teeth with exposed cervical dentin up to 1 mm deep and/or class I gingival recession according to the Miller classification;
* individuals who have at least two hypersensitive teeth
* periodontal health,
* good general physical health;
* willingness to participate in the research by providing written informed consent;
* no eating disorders or very acidic diets

Exclusion Criteria:

* presence of restorations;
* presence of dental caries and periodontal pockets;
* ongoing treatment with antibiotics and/or anti-inflammatory and/or analgesic drugs;
* professional desensitizing treatment received three months prior to the study;
* pregnancy or lactation; systemic diseases;
* pulpitis;
* use of orthodontic appliances or dental prostheses that may interfere with the assessment of hypersensitivity

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
sensitivity assessment | 30 days
  Evaluation of hypersensitivity in teeth with non-carious cervical lesions. Patients will be instructed to complete a form to record tooth sensitivity before the application of the gels. An evaluation will be performed at baseline, 7 days, 15 days and 30 days, based on their individual perception of pain. The evaluation form will consist of a visual analogue scale (VAS). This scale consists of a 10 cm horizontal line with points of 0 and 10 at its ends, where 0 means no sensitivity and 10 means severe tooth sensitivity. The patient will be instructed to draw a vertical line along the horizontal line of the scale, recording the intensity of tooth sensitivity. So that the distance in millimeters from the zero end can later be measured with the aid of a millimeter ruler, thus obtaining the intensity level of the patient's back.

CONTACTS AND LOCATIONS:
Overall Officials: Cecy M Silva, Doctor, Principal Investigator — universidade federal do pará
Locations (1):
- Universidade Federal Do Para, Belém, Pará, Brazil